CLINICAL TRIAL: NCT05812027
Title: Screening Study to Determine HLA Type, HLA Loss of Heterozygosity Status and Tumor Antigen Expression in Participants With Locally Advanced (Unresectable) or Metastatic Solid Tumors
Brief Title: A Screening Study to Collect Samples for TAA, HLA & HLA Loss of Heterozygosity in Patients With Metastatic Solid Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TSCAN-003
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer; Cervical Cancer; Non Small Cell Lung Cancer; HPV16 Related Cancers; Sarcoma; Uveal Melanoma; NUT Carcinoma
Keywords: Loss of Heterozygosity; HLA; Carcinoma; MAGE-A1; Adenocarcinoma; Squamous Cell Carcinoma; Epithelial Carcinoma; HPV Positive Cancers; TScan Therapeutics; TSCAN-002; TSCAN-003; PRAME; MAGE-C2; MAGE-A4; Sarcoma; Human Papillomavirus; Solid Tumor; HPV Positive Anogenital Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Sarcoma; Uveal Melanoma; Carcinoma; Adenocarcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Diagnostic Test: Tumor Profiling for TAA expression, HLA typing and HLA loss.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tumor and HLA Profiling — HLA genotyping and tumor tissue profiling for certain tumor-associated antigens and HLA LOH.

SUMMARY:
TScan Therapeutics is developing cellular therapies across multiple solid tumors in which autologous T cells are engineered to express a T cell receptor that recognizes tumor-associated antigens presented on specific Human Leukocyte Antigen (HLA) molecules. The purpose of this screening study is to collect samples to conduct HLA genotyping, HLA Loss of Heterozygosity (LOH) assessment, and expression of Tumor-associated Antigens (TAA) testing. These results will be used to determine if participants meet the eligibility criteria for these parameters and could potentially be enrolled in a TScan clinical study.

DETAILED DESCRIPTION:
This multicenter screening study will be conducted to determine a participant's tumor-associated antigen expression, HLA types and loss of HLA heterozygosity status for potential enrollment in a TScan sponsored clinical study. No treatment intervention will occur as part of this screening study.

Participants will be required to provide a buccal swab to assess their HLA types and a saliva sample to assess for HLA loss of heterozygosity. For participants with an HLA type for which TScan has an open clinical study, archival tissue (less than 8 months old) will be needed to assess for tumor-associated antigen expression. If archival tissue is not available or older than 8 months, a fresh tumor biopsy will be required.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Male or female aged ≥18 years at the time of signing the informed consent.
* Have one of the following histologically or cytologically confirmed locally advanced (unresectable) or metastatic solid tumor for which the Sponsor has an associated clinical study:
* Head and neck cancer
* Cervical cancer
* Non-small cell lung cancer
* HPV positive anogenital cancers
* Sarcoma
* Other cancers with a reasonable likelihood of expressing 1 or more antigens included in a TScan clinical trial, following approval by the TScan Medical Monitor or their delegate.
* Willing to provide a buccal swab for HLA testing
* Willing to provide a saliva sample to use as a normal control for the LOH assay
* Have access to an adequate FFPE tumor block that is <8 months old or is willing to provide a fresh core-needle biopsy from a location deemed safe by the treating medical team.

Exclusion Criteria:

• Participants undergoing anticancer therapy with curative intent such as tumor surgical resection with or without neoadjuvant/adjuvant therapy, or definitive chemoradiation, unless they have locoregionally advanced disease and are expected to have a high risk of relapse after their curative intent therapy as determined by the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to identify participants with locally advanced (unresectable) or metastatic solid tumors that could potentially be eligible for a TScan clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Frequency of subjects with TAA expression, HLA typing and HLA loss. | 3 years
  To identify participants that could potentially be eligible for the TScan Therapeutics clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Pinchasik, MD, Study Director — TScan Therapeutics, Inc.
Locations (21):
- United States (21):
  - HonorHealth Research and Innovation Institute, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Healthcare System, Hollywood, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Allegheny Hospitals Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided